CLINICAL TRIAL: NCT03423472
Title: Evaluation of Orange Fleshed Sweet Potato Promotion and the Healthy Baby Toolkit in Southern Ethiopia: a Cluster Randomized Controlled Trial
Brief Title: Improving Infant Nutrition in Southern Ethiopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Amy Webb Girard, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00099964
Record Dates: First submitted 2017-12-20; First posted 2018-02-06 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Nutrition Disorders
Keywords: Nutrition; Women; Young children; Ethiopia; Vitamin A; Orange flesh sweet potato
MeSH Terms: conditions — Nutrition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Full intervention (Experimental): Healthy Baby Toolkit (HBT) in addition to Orange Fleshed Sweet Potato (OFSP) agriculture promotion and education on family nutrition, with special emphasis on women and children < 2y; especially diet diversity and vitamin A intake
  Interventions: Behavioral: Orange Fleshed Sweet Potato (OFSP) agriculture promotion and nutrition education on vitamin A intake; Behavioral: Healthy Baby Toolkit; Behavioral: Standart of care
- Partial intervention (Active Comparator): Orange Fleshed Sweet Potato (OFSP) agriculture promotion and education on family nutrition, with special emphasis on women and children < 2y; especially diet diversity and vitamin A intake
  Interventions: Behavioral: Orange Fleshed Sweet Potato (OFSP) agriculture promotion and nutrition education on vitamin A intake; Behavioral: Standart of care
- Control (Other): Government standard of care for nutrition education through the Health Development Army
  Interventions: Behavioral: Standart of care

INTERVENTIONS:
Behavioral: Orange Fleshed Sweet Potato (OFSP) agriculture promotion and nutrition education on vitamin A intake — Support to farmers to grow and store OFSP in the form of agricultural extension, community based trainings and supplies, while simultaneously increasing community demand for OFSP through community-based Healthy Living Clubs. The Clubs promote OFSP, provide nutrition education, and conduct community mobilization events and social marketing of OFSP and OFSP-based processed products. Special emphasis is on women and children < 2y; especially diet diversity and vitamin A intake.
  Arms: Full intervention; Partial intervention
Behavioral: Healthy Baby Toolkit — The toolkit consists of a demarcated bowl, a slotted spoon, and a counseling card. The demarcations on the bowl guide caregivers on age-specific meal volume and frequency. The slotted spoon promotes thicker food consistency - and therefore nutrient density - by cuing caregivers when food drips through the slots. The counseling card relies on images rather than text to reinforce messages of the previous two instruments, promote dietary diversity, and promote hygienic food preparation.
  Arms: Full intervention
Behavioral: Standart of care — Government standard of care for nutrition education through the Health Development Army

SUMMARY:
This cluster randomized controlled trial will test the effect of the promotion of vitamin A-rich orange flesh sweet potato (OFSP) production and nutrition education on vitamin A and energy intake, including any added value of the Healthy Baby Toolkit.

DETAILED DESCRIPTION:
Child stunting and vitamin A deficiency are persistent public health problems in Ethiopia.

Quality Diets for Better Health (QDBH) is a European Union-funded project led by the International Potato Center (CIP), in partnership with People in Need (PIN), Emory University and with support of governmental organizations and local universities. The 54 month-project strives to improve diet quality, primarily of women and young children, through the promotion of vitamin A-rich orange flesh sweetpotato (OFSP) production and nutrition education in 41 kebeles (communities) in SNNPR, reaching an estimated 15000 households. In addition, households in a subset of communities will receive a Healthy Baby Toolkit, consisting of a marked bowl, slotted spoon, and illustrated counseling card. The Healthy Baby Toolkit is designed to promote optimal complementary feeding practices of infants and young children 6 to 23 months, namely meal volume, meal frequency, and meal thickness.

As part of this project, Emory University will conduct a longitudinal, cluster randomized controlled trial in 20 kebeles to test the effect of the project on vitamin A and energy intake, including any added value of the Healthy Baby Toolkit.

ELIGIBILITY:
Inclusion Criteria:

1. Participation in a Healthy Living Club (only a criteria for those in partial or full intervention arms)
2. Infant aged birth to 5 months
3. Primary caregiver and head of household (if different from primary caregiver) available and provides consent for survey

Exclusion Criteria:

1. Serious health problem (for example, HIV/AIDS or congenital defect)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 605 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Change in vitamin A intake of young children | Baseline, approximately 6 months at midline, and approximately 1 year at endline
  Multiple linear regression will be used to explore the effect of intervention status on vitamin A intake, while controlling for covariates and assessing interaction. The Ethiopian Food Composition Tables I-IV will be used to derive the data from dietary data collected at midline and at endline.
Change in energy intake of young children | Baseline, approximately 6 months at midline, and approximately 1 year at endline
  Multiple linear regression will be used to explore the effect of intervention status on energy intake, while controlling for covariates and assessing interaction. The Ethiopian Food Composition Tables I-IV will be used to derive the data from dietary data collected at midline and at endline.

SECONDARY OUTCOMES:
Validation of survey-based indicators of meal volume for children ages 6 to 11 months | Approximately 6 months at midline, and approximately 1 year at endline
  Nutrient intake data collected at midline and endline will be compared with caregiver responses to indicator questions using combinations of the following: Bland Altman plots, Pearson's correlation, sensitivity and specificity, and/or Receiver Operating Characteristic Curves.
Validation of survey-based indicators of food consistency for children ages 6 to 11 months | Approximately 6 months at midline, and approximately 1 year at endline
  Nutrient density data collected at midline and endline will be compared with caregiver responses to indicator questions using combinations of the following: Bland Altman plots, Pearson's correlation, sensitivity and specificity, and/or Receiver Operating Characteristic Curves.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Girard, Principal Investigator — Emory University
Locations (2):
- Emory University, Atlanta, Georgia, United States
- International Potato Center (CIP), Sīdamo, Southern Nations, Nationalities, and Peoples' Region (snnpr), Ethiopia